CLINICAL TRIAL: NCT03065543
Title: Hyperlipidemia Therapy in tERtiary Cardiological cEnTer Zabrze Registry
Brief Title: Hyperlipidemia Therapy TERCET Zabrze Registry
Acronym: TERCETZabrze
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Prof. of Medicine, Head of 3rd Department of Cardiology, SMDZ in Zabrze, Medical University of Silesia, Katowice, Poland, Silesian Centre for Heart Diseases
Other Study IDs: III KOK 01/2017
Record Dates: First submitted 2017-02-07; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Hyperlipidemias; Secondary Prevention
Keywords: Hyperlipidemias; Secondary prevention; high risk patients; very high risk patients
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A study conducted to evaluate the efficacy of lipid-lowering therapy in patients with high and very high risk treated by interventional cardiology. Study endpoints:

1. Achievement of the target LDL-C at 1-year follow-up LDL-C <70 mg / dl in the group of very high-risk and LDL-C <100 mg / dL in high-risk patients
2. Assessment of the lipid profile of the severity of coronary artery disease in patients undergoing invasive diagnosis of coronary artery disease
3. Evaluation of trends in the treatment of lipid-lowering in patients in different years

DETAILED DESCRIPTION:
The TERCET Zabrze Registry is an observational study of all patients hospitalized due to the cardiovascular diseases. The date include information on the hyperlipidaemia treatment, clinical characteristics, any treatment modalities and prognosis in this population. Data collection is patient-based (not event-based).

The study population is formed by all-comer patients hospitalized in cardiology wards and intensive cardiac care units with a diagnosis of coronary disease, both stable angina, and acute coronary syndromes (ACS). For the purpose of this study hyperlipidaemia is defined in accordance with European Society of Cardiology guidelines.

Complete patient demographics; medical history, complete hospitalization data (diagnostic and therapeutic), in-hospital and out-hospital results are collected in an electronic form by the attending physician. The patients are under constant follow-up for all cause mortality and major adverse events.

ELIGIBILITY:
Inclusion Criteria:

* All patients with coronary artery disease with hyperlipidemia

Exclusion Criteria:

* No coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is formed by all patients hospitalized in the 3-Dept of Cardiology Zabrze, Poland due to cardiovascular diseases and hyperlipidemia from 1st January 2006.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of treatment on the lipid profile and long-term prognosis | 2006-2025
  The registry compares lipid profile values (assayed by the standard laboratory techniques): total cholesterol (TCh), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), and TG (triglycerides) with an intense emphasis on the LDL-C value measured during the inclusion to the registry, with MACE (Major Adverse Cardiac Events) and a control lipid profile measurement, depending on the therapy form (revascularization followed by an intensified pharmacological treatment/revascularization only/pharmacological treatment only). The information regarding MACE is acquired from the NFZ (National Health Fund; polish healthcare provider). Using the statistical analysis the influence of an optimised hyperlipidemia treatment on the long-term prognosis will be assessed.

SECONDARY OUTCOMES:
Assessment of the lipid profile of the severity of coronary artery disease | 2006-2025
  A comparison of an initial lipid profile values (with an intense emphasis on the LDL-C), assayed by the standard laboratory techniques) and the coronary artery atherosclerosis extensity, and the long-term prognosis in a year after discharge from hospital. The information regarding MACE is acquired from the NFZ (National Health Fund; polish healthcare provider). Using the statistical analysis the influence of an optimised hyperlipidemia treatment on the long-term prognosis will be assessed.
Evaluation of trends in the treatment of lipid-lowering in patients in different years | 2006-2025
  An observation of TCh, LDL-C, HDL-C and TG serum concentration values (measured by the standard laboratory assay techniques) depending on the period of the Registry function and the date of inclusion to the Registry. This part of the examination will answer how do the physicians adhere to the hyperlipidemia treatment guidelines in Poland and what are the trends in this therapy form.

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Gasior, prof.MD,PhD, Principal Investigator — 3rd Department of Cardiology, SMDZ in Zabrze, Medical University of Silesia, Katowice, Poland
Locations (1):
- Silesian Center for Heart Diseases, Zabrze, Upper Silesia, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dyrbus K, Osadnik T, Desperak P, Desperak A, Gasior M, Banach M. Evaluation of dyslipidaemia and the impact of hypolipidemic therapy on prognosis in high and very high risk patients through the Hyperlipidaemia Therapy in tERtiary Cardiological cEnTer (TERCET) Registry. Pharmacol Res. 2018 Jun;132:204-210. doi: 10.1016/j.phrs.2017.12.015. Epub 2017 Dec 16. PMID 29258913